CLINICAL TRIAL: NCT06799546
Title: A Phase III, Multicenter, Randomized, Open Label, Active-Controlled Study to Evaluate the Efficacy and Safety of HSK39297 Tablets in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH) Who Are Naive to Complement Inhibitor Therapy
Brief Title: A Phase III Study to Evaluate the Efficacy and Safety of HSK39297 in Patients With Paroxysmal Nocturnal Hemoglobinuria Who Are Naive to Complement Inhibitor Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK39297-301
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: PNH
MeSH Terms: interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK39297 tablets (Experimental)
  Interventions: Drug: HSK39297 tablets
- Eculizumab Injection (Active Comparator)
  Interventions: Drug: Eculizumab Injection

INTERVENTIONS:
Drug: HSK39297 tablets — 200mg QD for 24 weeks
  Arms: HSK39297 tablets
Drug: Eculizumab Injection — Eculizumab Injection for 24 weeks
  Arms: Eculizumab Injection

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of HSK39297 tablets compared to eculizumab in Patients with PNH who Are Naive to Complement Inhibitor Therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years, Male and female patients;
2. Diagnosis of PNH based on flow cytometry with clone size > 10% by granulocytes;
3. Have not received complement inhibitor treatment;
4. Blood LDH values > 1.5 ×upper limit of the normal range (ULN) ;
5. Hemoglobin level < 10 g/dL at screening.

Exclusion Criteria:

1. Hereditary or acquired complement deficiency;
2. Active primary or secondary immunodeficiency;
3. History of splenectomy, bone marrow/ hematopoietic stem cell or solid organ transplants;
4. History of recurrent invasive infections caused by encapsulated organisms( e.g. meningococcus or pneumococcus) or Mycobacterium tuberculosis;
5. Patients with laboratory evidence of bone marrow failure (reticulocytes < 100x10^9/L, or platelets < 30x10^9/L or neutrophils < 0.5x10^9/L) ;
6. Active systemic infection within 2 weeks prior to study drug administration;
7. History of serious comorbidities that have been determined to be unsuitable for participation in the study.
8. Pregnant or Lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving hemoglobin levels ≥ 12 g/dL at least on three out of four measurements in the absence of red blood cell transfusions | Between Week 18 and Week 24

SECONDARY OUTCOMES:
Proportion of participants with increase in hemoglobin levels from baseline of ≥20 g/L at least on three out of four measurements in the absence of red blood cell transfusions | Between Week 18 and Week 24
Proportion of participants who did not receive blood transfusion. | Between Week 2 and Week 24
Change from baseline in hemoglobin | Baseline, week 18 to 24
Change From Baseline in Reticulocyte Count | Baseline, week 18 to 24
Percent change from baseline in LDH | Baseline, week 18 to 24
Change from baseline in FACIT-Fatigue score | Baseline, week 18 to 24
Rate of breakthrough hemolysis (BTH) | 24 weeks
Proportion of participants with Major Adverse Vascular Events (MAVEs) | 24 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided